CLINICAL TRIAL: NCT02903160
Title: Clinical Trial of a Rapidly Cycling, Non-Cross Reactive Regimen of Approved Therapeutic Agents to Treat Prostate Cancer
Brief Title: Prostate Cancer Intensive, Non-Cross Reactive Therapy (PRINT) for Castration Resistant Prostate Cancer (CRPC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Sanofi (Industry); Bayer (Industry)
Responsible Party: Principal Investigator, Bobby Liaw, Assistant Profesor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 16-1593; CABAZL07459 (Other: Sanofi); ONC-2014-168 (Other: Bayer)
Record Dates: First submitted 2016-09-07; First posted 2016-09-16 (Estimated); Results first posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer
Keywords: Castration resistant; Prostate cancer; Metastatic; First-line; Treatment naive; Rapidly cycling; Non-cross resistant
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — Abiraterone Acetate; Prednisone; radium Ra 223 dichloride; cabazitaxel; Carboplatin; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intensive, Non-Cross Reactive Therapy (Experimental): Prostate Cancer Rapidly cycling, Intensive, Non-Cross Reactive Therapy (PRINT) Rapidly cycling, consecutive treatment modules: 1. Abiraterone acetate; 2. Cabazitaxel + Carboplatin; 3. Enzalutamide + Radium-223
  Interventions: Drug: Abiraterone acetate; Drug: Prednisone; Drug: Radium-223 dichloride; Drug: cabazitaxel; Drug: Carboplatin; Drug: Enzalutamide

INTERVENTIONS:
Drug: Abiraterone acetate — Abiraterone acetate 1000 mg PO daily
Drug: Prednisone — 5 mg PO twice a day
Drug: Radium-223 dichloride — 50 kBq/kg IV monthly
Drug: cabazitaxel — 25 mg/m2 IV every 3 weeks
Drug: Carboplatin — Carboplatin AUC 4 IV every 3 weeks
Drug: Enzalutamide — 160 mg PO daily

SUMMARY:
The purpose of this study is to determine the clinical benefits of using a rapidly cycling, non-cross reactive regimen of FDA-approved prostate cancer therapeutic agents in the management of castration resistant prostate cancer. The hypothesis is that the identification of optimal combinations and sequencing of therapies can help prevent or delay the development of therapeutic drug resistance, and can be safely tolerated.

DETAILED DESCRIPTION:
This phase II clinical trial will explore the efficacy of rapidly cycling non-cross reactive treatment therapies in the treatment of patients with newly diagnosed mCRPC. The primary hypothesis is that the best chance of eliminating or controlling disease is when the cancer is treatment naïve, and has not yet developed therapeutic resistance. By finding an optimal drug deployment strategy of already approved and available treatments for mCRPC, the researchers believe providers can more effectively treat an intrinsically heterogeneous disease, delay/prevent drug resistance, as well as minimize treatment toxicity.

All of the treatment agents selected have well-defined individual toxicity profiles from large phase III trials, but there is limited clinical data about the toxicity profiles of these drugs in combinations. While each agent is generally well tolerated, toxicities remain a significant concern given the older age of the typical mCRPC patient, the comorbid conditions common to this patient population, as well as those borne from previous chronic androgen deprivation therapy.

Each drug in the proposed treatment regimen will be used at their FDA-approved dosing and indication, with the exception of cabazitaxel, which will be used prior to disease demonstration of docetaxel failure, and in combination with carboplatin. The proposed sequencing is rationally designed, and based on each drug's distinct mechanisms of action as well as their toxicity profiles.

The rapidly-cycling treatment regimen contains three, separate, consecutive treatment modules, each lasting 3 months: 1. Abiraterone; 2. Cabazitaxel + Carboplatin; 3. Enzalutamide + Radium-223. Therapeutic agents are delivered as non-cross reactive combinations, in order to achieve optimal therapeutic dosing at each cycle and decrease possibility of significant adverse effects.

To the researcher knowledge, no study has evaluated the use of rapidly cycling, non-cross reactive therapies for the treatment of mCRPC. The hypothesis is that the identification of optimal combinations and sequencing of rapidly cycling non-cross reactive therapies can help prevent or delay the development of therapeutic drug resistance, and can be safely tolerated.

Primary objective is to evaluate the time to disease progression after completion of all modules of the rapidly-cycling, non-cross reactive regimen in patients with mCRPC. Secondary objectives are to evaluate overall survival, prostate-specific antigen (PSA) response rate with each treatment module, changes to alkaline phosphatase level, and assess safety of the rapidly-cycling, non-cross reactive regimen. Additional exploratory objective are to evaluate the correlation of a peripheral whole-blood RNA signature with clinical outcome measures during and after treatment, and to evaluate changes to AR-V7 expression in CTCs with different treatment modalities and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate
* Metastatic castrate resistant prostate cancer, defined by progressive disease based on either rising PSA, new bone metastases, or progression of measurable disease on standard imaging, according to PCWG2 guidelines, despite androgen deprivation therapy
* Ongoing androgen deprivation therapy with a GnRH analogue, GnRH antagonist, or bilateral orchiectomy
* ECOG performance status 0-1
* Serum testosterone level < 50 ng/dL
* Absolute neutrophil count > 1,500/μL, platelet count > 100,000/μL, and hemoglobin > 9 g/dL
* Creatinine < 2 mg/dL
* Total bilirubin < 1 times the upper limit of normal, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 1.5 times the upper limit of normal

Exclusion Criteria:

* History of uncontrolled seizure disorder
* Clinically significant cardiovascular disease including:

  1. Myocardial infarction or uncontrolled angina within 6 months
  2. Congestive heart failure New York Heart Association (NYHA) class 3 or 4, or patients with history of congestive heart failure NYHA class 3 or 4 in the past
  3. Uncontrolled hypertension as indicated by a resting systolic blood pressure > 170 mmHg or diastolic blood pressure > 105 mmHg at the screening visit
* Have used or plan to use from 30 days prior to enrollment through the end of the study medication known to lower the seizure threshold or prolong the QT interval
* Major surgery within 4 weeks of enrollment
* Radiation therapy within 4 weeks of enrollment
* Prior use of abiraterone acetate, enzalutamide, docetaxel, cabazitaxel, carboplatin, or radium-223 for the treatment of castration-resistant disease
* Prior docetaxel use in the hormone-sensitive disease setting is allowed, but must be completed ≥ 4 weeks prior to enrollment
* Prior sipuleucel-T use is allowed, but must be completed ≥ 4 weeks prior to enrollment
* Concurrent use of zoledronic acid or denosumab is allowed on study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bobby Liaw, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Mount Sinai Beth Israel, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intensive, Non-Cross Reactive Therapy: Prostate Cancer Rapidly cycling, Intensive, Non-Cross Reactive Therapy (PRINT) Rapidly cycling, consecutive treatment modules: 1. Abiraterone acetate 1000 mg PO daily; 2. Cabazitaxel 25 mg/m2 IV every 3 weeks + Carboplatin AUC 4 IV every 3 weeks; 3. Enzalutamide 160 mg PO daily + Radium-223 kg IV monthly and Prednisone: 5 mg PO twice a day
Period: Overall Study
Arm/Group | Intensive, Non-Cross Reactive Therapy
Started | 40
Completed | 33
Not Completed | 7
Not completed — Adverse Event | 2
Not completed — Death | 1
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 1
Not completed — Medical Insurance Barriers | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intensive, Non-Cross Reactive Therapy
Number analyzed (Participants) | 40
Age, Continuous [Mean (Full Range); unit: years] | 69 [48 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Amerian Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 21
  Hispanic | 7
  More than one race | 0
  Unknown or Not Reported | 1
Gleason score [Count of Participants; unit: Participants] — Gleason scores ranges from 2-10. A score of 6 is low grade, 7 is intermediate grade, and a score of 8 to 10 is high grade cancer.
  Participants
    <=6 | 5
    7 | 10
    >=8 | 21
    Unknown | 4
Prostate-specific antigen (PSA) [Median (Inter-Quartile Range); unit: ng/mL] | 9.6 [4.8 to 40.3]
Alkaline phosphatase [Median (Inter-Quartile Range); unit: IU/L] | 98 [77.8 to 153]
Alkaline phosphatase [Count of Participants; unit: Participants]
  Elevated (>126 IU/L) | 13
  Normal (<=126 IU/L) | 27
Eastern Cooperative Oncology Group (ECOG) [Count of Participants; unit: Participants] — ECOG Performance Status Scale:
  0 Fully active, able to carry on all pre-disease performance without restriction
  1 Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  Participants
    0 | 27
    1 | 10
    unknown | 3
Sites of metastasis [Count of Participants; unit: Participants]
  Bone | 29
  Lymph node | 13
  Lung | 1
  Liver | 0
  Other | 2

OUTCOME MEASURES:

1. Primary Outcome: Time to Disease Progression
Description: Time to disease progression, as determined by either PSA or radiographic progression, after completion of all modules of the rapidly-cycling, non-cross reactive regimen in patients with mCRPC.
  Time to progression (TTP) is defined as beginning with the time the first dose of PCD regimen is administered until disease progression.
Time Frame: 47.8 months
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Intensive, Non-Cross Reactive Therapy
Number analyzed (Participants) | 33
weeks | 15.2 [10.8 to 23.2]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival defined as the time of study entry to death from any cause.
Time Frame: 47.8 months
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Intensive, Non-Cross Reactive Therapy
Number analyzed (Participants) | 33
weeks | NA [NA to NA] — Median OS not reached. Not enough events that have occurred to have a median OS. Not enough event data to estimate the lower and the upper bound of the 95% CI for median OS.

3. Secondary Outcome: Overall Rate of Survival
Description: Overall rate of survival at 40 months. Overall rate of Survival as defined by likelihood that a participant on the study is still alive at 40 months follow up
Time Frame: 40 months
Measure: Median (95% Confidence Interval); unit: percent
Arm/Group | Intensive, Non-Cross Reactive Therapy
Number analyzed (Participants) | 33
percent | 63 [47 to 85]

4. Secondary Outcome: Number of Participants With PSA Response Rate >90%
Description: PSA response rate - >90% decrease in PSA compared to baseline
Time Frame: up to 36 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive, Non-Cross Reactive Therapy
Number analyzed (Participants) | 33
Participants
  after module 1, 12 weeks | 11
  after module 2, 24 weeks | 14
  after module 3, 36 weeks | 20

5. Secondary Outcome: Number of Participants With PSA Response Rate >=50%
Description: Number of participants with PSA response rate >=50% decrease in PSA compared to baseline
Time Frame: up to 36 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive, Non-Cross Reactive Therapy
Number analyzed (Participants) | 33
Participants
  after module 1, 12 weeks | 27
  after module 2, 24 weeks | 28
  after module 3, 36 weeks | 32

6. Secondary Outcome: Number of Participants With PSA Progression Compared to Baseline.
Description: PSA changes was reported globally using a waterfall plot for each module. In participants who have a decline in PSA value from baseline, progression is defined by:
  * An increase in PSA by 25% above the nadir, AND
  * An increase in PSA by a minimum of 2 ng/ml, or an increase in PSA to the pre-treatment PSA value, AND
  * Confirmation by a second PSA at least 3 weeks apart, AND
  * Occur following at least 12 weeks of therapy, AND
  * There is no objective evidence of disease response.
  In participants whose PSA value from baseline has not declined from baseline, progression is defined by:
  * An increase in PSA by 25% above either the pre-treatment level, or the nadir PSA level (whichever is lowest), AND
  * An increase in PSA by a minimum of 2 ng/ml, AND
  * Confirmation by a second PSA at least 3 weeks apart, AND
  * Occur following at least 12 weeks of therapy, AND
  * There is no objective evidence of disease response.
Time Frame: up to 36 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive, Non-Cross Reactive Therapy
Number analyzed (Participants) | 33
Participants
  after module 1, 12 weeks | 4
  after module 2, 24 weeks | 4
  after module 3, 36 weeks | 0

7. Secondary Outcome: Number of Participants With Stable PSA as Compared to Baseline
Description: Participants with a 50% PSA decline from their baseline PSA level will be considered responders, provided objective tumor measurements are stable or also demonstrate response. Participants with a 25% PSA increase from their baseline PSA will be considered nonresponders. Participants that do not meet criteria for responder or nonresponder, will be considered to have stable disease.
Time Frame: up to 36 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive, Non-Cross Reactive Therapy
Number analyzed (Participants) | 33
Participants
  after module 1, 12 weeks | 2
  after module 2, 24 weeks | 1
  after module 3, 36 weeks | 1

8. Secondary Outcome: Number of Participants With Normal Alkaline Phosphatase Levels
Description: Number of participants who converted from elevated to normal range of alkaline phosphatase levels at 9 months from baseline
Time Frame: baseline and 36 weeks
Population: Data for those with elevated alkaline phosphatase levels at baseline and with results available at 36 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive, Non-Cross Reactive Therapy
Number analyzed (Participants) | 10
Participants | 8

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from enrollment up to 48 weeks. All-Cause Mortality was from first dose until death, assessed up to 47.8 months
Arm/Group | Intensive, Non-Cross Reactive Therapy
All-Cause Mortality (participants affected / at risk) | 1/33
Serious Adverse Events (participants affected / at risk) | 10/33
Other Adverse Events (participants affected / at risk) | 18/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intensive, Non-Cross Reactive Therapy (N=33)
hyperglycemia (Endocrine disorders) | 1
vomiting (Gastrointestinal disorders) | 1
diarrhea (Gastrointestinal disorders) | 2
nausea (Gastrointestinal disorders) | 1
lymphocyte count decreased (Blood and lymphatic system disorders) | 1
platelet count decreased (Blood and lymphatic system disorders) | 1
neutrophil count decreased (Blood and lymphatic system disorders) | 2
blood bilirubin increased (Hepatobiliary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intensive, Non-Cross Reactive Therapy (N=33)
hyperglycemia (Endocrine disorders) | 7
vomiting (Gastrointestinal disorders) | 9
diarrhea (Gastrointestinal disorders) | 17
nausea (Gastrointestinal disorders) | 14
lymphocyte count decreased (Blood and lymphatic system disorders) | 13
platelet count decreased (Blood and lymphatic system disorders) | 6
neutrophil count decreased (Blood and lymphatic system disorders) | 5
fatigue (General disorders) | 18
white blood cell count decreased (Blood and lymphatic system disorders) | 13
anorexia (Gastrointestinal disorders) | 13
anemia (Blood and lymphatic system disorders) | 13
hypertension (Cardiac disorders) | 3
alanine aminotransferase increased (Hepatobiliary disorders) | 4
aspartate aminotransferase increased (Hepatobiliary disorders) | 5
arthralgia (Musculoskeletal and connective tissue disorders) | 2
atrial flutter (Cardiac disorders) | 1
bloating (Gastrointestinal disorders) | 2
constipation (Gastrointestinal disorders) | 2
creatinine increased (Renal and urinary disorders) | 1
dizziness (Nervous system disorders) | 3
dysgeusia (Gastrointestinal disorders) | 5
dyspepsia (Gastrointestinal disorders) | 1
dysphagia (Gastrointestinal disorders) | 1
dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
edema limbs (Vascular disorders) | 2
hot flashes (Endocrine disorders) | 6
flu like symptoms (Immune system disorders) | 1
gastroesophageal reflux disease (Gastrointestinal disorders) | 1
hypoalbuminemia (Hepatobiliary disorders) | 1
hypokalemia (Renal and urinary disorders) | 1
hypotension (Cardiac disorders) | 1
infusion related reaction (General disorders) | 1
blood lactate dehydrogenase increased (General disorders) | 1
muscle cramp (Musculoskeletal and connective tissue disorders) | 1
muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
malaise (General disorders) | 1
generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
bone pain (Musculoskeletal and connective tissue disorders) | 2
hyperhydrosis (Endocrine disorders) | 1
peripheral motor neuropathy (Nervous system disorders) | 1
peripheral sensory neuropathy (Nervous system disorders) | 10
phlebitis (Vascular disorders) | 1
maculopapular rash (Skin and subcutaneous tissue disorders) | 1
skin infection (Skin and subcutaneous tissue disorders) | 1
urinary tract pain (Renal and urinary disorders) | 1
abdominal pain (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/60/NCT02903160/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/60/NCT02903160/ICF_001.pdf